CLINICAL TRIAL: NCT06630078
Title: Artificial Intelligence-based Voice Assessment of Children and Adults With Acute and Chronic Respiratory Conditions: Diagnostic and Prognostic Role
Brief Title: Artificial Intelligence-based Voice Assessment of Children and Adults Respiratory Conditions
Acronym: AIRWAY-VDAP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Galli Jacopo, Full Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ID6812
Record Dates: First submitted 2024-07-25; First posted 2024-10-08 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Airway Disease; Cancer of Head and Neck; Radiotherapy; Bronchiolitis; Asthma
MeSH Terms: conditions — Head and Neck Neoplasms; Bronchiolitis; Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Case group (Experimental): children with bronchiolits, controlled asthma and asthmatic re-exacerbations and adults with primary upper aero-digestive tract affections or secondary to radiotherapy
  Interventions: Device: Wevosys acoustic analysis

INTERVENTIONS:
Device: Wevosys acoustic analysis — Recording of voice signal of subjects enrolled

SUMMARY:
Acute and Chronic respiratory conditions represent a leading cause of death and morbidity in children and adults worldwide. The diagnosis of bronchiolitis and asthmatic exacerbations is based on clinical, and mostly subjective, clinical parameters with moderately accurate prognostic role. Patients undergoing neck radiotherapy need invasive assessments of larynx. A simple biomarker like Voice may facilitate the management of these conditions. Recent studies showed that VOICE may be used as a good and easy biomarker to diagnose and monitor several respiratory and non-respiratory conditions. A prospective study aimed to collected VOICE and other clinical data in adults and children with common acute and chronic respiratory conditions at high impact on healthcare systems will be performed. VOICE-omic data will be linked with clinical findings generating data integration, using artificial intelligence technology to develop a Decision Support Systems to provide the basis for non-invasive personalised early recognition, diagnosis, monitoring and prognosis of patients with these conditions.

ELIGIBILITY:
INCLUSION CRITERIA:

* Children with bronchiolitis <24 months of age clinically characterized according to the clinical definition accepted by international literature (Ralstone);
* Children with asthma according to most recent GINA guidance (Global Initiative for Asthma, 2022) aged 6-12 years in a phase of proper control or during acute exacerbations;
* Adults with upper aerodigestive tract chronic or acute clinical conditions;
* Adults with pathologic diagnosis of head and neck cancer addressed to radiotherapy with or without chemotherapy for primary treatment of the tumor.

EXCLUSION CRITERIA:

* Children with comorbidities including genetic disorders;
* Children with other chronic respiratory conditions (bronchodysplasia, cystic fibrosis);
* Children with primary immunologic diseases;
* Children with prematurity;
* Children with other respiratory conditions not part of the inclusion criteria (examples: pneumonia, tonsillitis);
* Adults over 70 years old or with neurological diseases;
* Adults with syndromic disease;
* Adults with malformations of upper aero-digestive tract;
* Adults with history of head and neck surgery or not able to sustain a vocalism for more than 3 sec.

Ages: 12 Months to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Acoustic parameters of voice signal in children | enrollment; 24 and 48 hours post-therapy; 24 months
  Fundamental frequency (F0), measured in Hertz, is defined as the number of times a sound wave produced by the vocal cords repeats during a given time period, it is also the number of cycles of opening/closure of the glottis.
Acoustic parameters of voice signal in children | enrollment; 24 and 48 hours post-therapy; 24 months
  Jitter (%) is the variation from cycle of opening/closure of the glottis to cycle.
Acoustic parameters of voice signal in children | enrollment; 24 and 48 hours post-therapy; 24 months
  Shimmer (%) relates to the amplitude variation of the sound wave.
Acoustic parameters of voice signal in children | enrollment; 24 and 48 hours post-therapy; 24 months
  NHR (decibel) that is an assessment of the ratio between periodic components and non periodic component comprising a segment of voiced speech.
Acoustic parameters of voice signal in adults affected by acute or chronic upper aerodigestive diseases | enrollment; 24 and 48 hours post-therapy; 24 months
  Fundamental frequency (F0), measured in Hertz, is defined as the number of times a sound wave produced by the vocal cords repeats during a given time period, it is also the number of cycles of opening/closure of the glottis.
Acoustic parameters of voice signal in adults affected by acute or chronic upper aerodigestive diseases | enrollment; 24 and 48 hours post-therapy; 24 months
  Jitter (%) is the variation from cycle of opening/closure of the glottis to cycle; Shimmer (%) relates to the amplitude variation of the sound wave.
Acoustic parameters of voice signal in adults affected by acute or chronic upper aerodigestive diseases | enrollment; 24 and 48 hours post-therapy; 24 months
  Shimmer (%) relates to the amplitude variation of the sound wave.
Acoustic parameters of voice signal in adults affected by acute or chronic upper aerodigestive diseases | enrollment; 24 and 48 hours post-therapy; 24 months
  NHR (decibel) that is an assessment of the ratio between periodic components and non periodic component comprising a segment of voiced speech.
Pediatric Dyspnea Scale | enrollment; 24 hours and 48 hours post-therapy; 24 months
  The child is asked to answer the question "How much difficulty are you having breathing?" by choosing the column that best corresponds to his or her perceived symptoms (range from 0 not trouble at all to 7 very much trouble)
Voice Handicap Index score in adults affected by acute or chronic upper aerodigestive diseases | enrollment; 24 hours and 48 hours after therapy; 24 months
  The Voice Handicap Index is self-assessment instrument useful for quantifying the biopsychosocial impact of a voice disorder. It consists of 30 items. The total score ranges from 0 (no impact of dysphonia) to 120 (the worst possibile impact of dysphonia)
Acoustic parameters of voice signal in adults underwent radiotherapy | enrollment; on the 30th day of radiotherapy
  Fundamental frequency (F0), measured in Hertz, is defined as the number of times a sound wave produced by the vocal cords repeats during a given time period, it is also the number of cycles of opening/closure of the glottis.
Acoustic parameters of voice signal in adults underwent radiotherapy | enrollment; on the 30th day of radiotherapy
  Jitter (%) is the variation from cycle of opening/closure of the glottis to cycle.
Acoustic parameters of voice signal in adults underwent radiotherapy | enrollment; on the 30th day of radiotherapy
  Shimmer (%) relates to the amplitude variation of the sound wave.
Acoustic parameters of voice signal in adults underwent radiotherapy | enrollment; on the 30th day of radiotherapy
  NHR (decibel) that is an assessment of the ratio between periodic components and non periodic component comprising a segment of voiced speech.
Voice Handicap Index score in adults who underwent radiotherapy | enrollment; on the 30th day of radiotherapy
  The Voice Handicap Index is self-assessment instrument useful for quantifying the biopsychosocial impact of a voice disorder. It consists of 30 items. The total score ranges from 0 (no impact of dysphonia) to 120 (the worst possibile impact of dysphonia)
Dysphagia Handicap Index in adults who underwent radiotherapy | enrollmentt; on the 30th day of radiotherapy
  The Dysphagia Handicap Index is a 25-item measure of Health-related Quality of Life for patients with oropharyngeal dysphagia of heterogeneous etiologies. The total score ranges from 0 to 100, with lower scores indicating better swallowing-related QoL.

CONTACTS AND LOCATIONS:
Overall Officials: Jacopo Galli, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (2):
- Italy (2):
  - Jacopo Galli, Roma
  - Maria Raffaella Marchese, Roma

IPD SHARING:
Plan to Share IPD: No